CLINICAL TRIAL: NCT07143318
Title: A Phase I Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Single and Multiple Doses of KLA578-1 for Injection in Healthy Volunteers
Brief Title: First-in-Human Single and Multiple Dose of KLA578-1 for Injection
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sichuan Kelun Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Organization: Sichuan Kelun Pharmaceutical Research Institute Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KLA578-1-101
Record Dates: First submitted 2025-07-23; First posted 2025-08-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-07

CONDITIONS: Healthy Volunteers
Keywords: Healthy
MeSH Terms: interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- KLA578-1 60mg (Experimental): 12 volunteers receive KLA578-1 for injection 60mg
  Interventions: Drug: KLA578-1 for injection
- KLA578-1 120mg (Active Comparator): Period 1, 6 volunteers receive KLA578-1 for injection 120mg → 6 volunteers receive Etopcoxib Tablets 120mg; Period 2, 6 volunteers receive Etopcoxib Tablets 120mg → 6 volunteers receive KLA578-1 for injection 120mg
  Interventions: Drug: KLA578-1 for injection; Drug: Etopcoxib Tablets
- KLA578-1 240mg (Experimental): 12 volunteers receive KLA578-1 for injection 240mg
  Interventions: Drug: KLA578-1 for injection
- multiple doses of KLA578-1 for injection (Experimental): 12 volunteers receive KLA578-1 for injection 120mg over 5 consecutive days.
  Interventions: Drug: KLA578-1 for injection

INTERVENTIONS:
Drug: KLA578-1 for injection — Intravenous injection, single dose
Drug: Etopcoxib Tablets — P.O., single dose
  Arms: KLA578-1 120mg

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability and pharmacokinetics of single and multiple doses of KLA578-1 for injection in healthy volunteers

DETAILED DESCRIPTION:
"The study will be carried out in 2 parts. Part 1: This is a open-label, single ascending dose (SAD) escalation study with a total of 3 dose groups, i.e., Groups 1 to 3. There are a total of 12 volunteers in each group with a similar male to female ratio. Groups 1 and 3 are single-arm study, all volunteers will receive the experimental drug ""KLA578-1 for Injection"" ; Group 2 is a randomized, two-treatment, two-period, crossover study, 12 volunteers will be randomized to TR sequence or RT sequence with 6 volunteers in each sequence. The experimental drug ""KLA578-1 for injection"" will be administered in the TR sequence of Period 1, the control drug ""Etopcoxib Tablets"" will be administered to the RT sequence. After 7 days of washing, the control drug ""Etocoxib Tablets"" will be administered in the TR sequence, and the experimental drug ""KLA578-1 for Injection"" will be administered in the RT sequence.

Part 2: This is a open-label, single-arm multiple dose study. A dose group is temporarily set up, with a total of 12 volunteers enrolled, and the male-to-female ratio will be similar. Volunteers will receive the experimental drug ""KLA578-1 for Injection"" 120 mg once daily (every 24 h ± 2 min with reference to the dosing time on D1) under fasting conditions (fasting for at least 10 hours) from D1 to D5; Drinking water is prohibited from 1 h before each dose to 1 h postdose, and fasted within 4 hours after dosing on D1 and D5."

ELIGIBILITY:
Inclusion Criteria:

1. Health Volunteers (Age: 18~45 years);
2. Body Weight: Male≥50.0kg, Female≥45.0kg; 19.0 ≤BMI≤ 26.0;
3. There were no abnormalities in clinically significant physical examination, vital signs, 12-lead electrocardiogram, laboratory tests;
4. Heart rate ≥ 60 bpm and pulse ≥ 60 beats/min.

Exclusion Criteria:

1. Allergy or Drug hypersensitivity;
2. Clinically significant Medical History;
3. Gastrointestinal ulcers or gastrointestinal bleeding;
4. History of any surgery within 4 weeks;
5. History of any Medication within 14 days;
6. History of any inducers or inhibitors of major CYP450 enzymes within 30 days;
7. History of any clinical study within 3 months;
8. History of any vaccine within 1 month;
9. History of any drug abuse;
10. Tablet dysphagia;
11. Needle sickness, Hematosickness;
12. Massive blood loss (> 200 mL) in the past 3 months;
13. Female volunteers are pregnant or lactating;
14. History of unprotected sex within 2 weeks;
15. Special requirements for diet;
16. Heavy smoker ( more than 3 cigarettes/day) within 3 months;
17. History of alcohol abuse,or heavy alcohol intake (more than 14 units a week) within 6 months;
18. Heavy caffeine intake;
19. History of grapefruit, xanthine-rich foods intake within 7 days;
20. Positive alcohol test;
21. Positive drugs of abuse test result.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-06-05 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events (AEs) | Up to day 13

SECONDARY OUTCOMES:
PK parameter Cmax | single dose：up to Day 6 ; multiple doses: up to Day 8
  Maximum peak plasma concentration (Cmax) after single dose and in a steady state after multiple doses
PK parameter Tmax | single dose：up to Day 6 ; multiple doses: up to Day 8
  Time of Cmax (Tmax) after single dose and in a steady state after multiple doses
PK parameter Cmin,ss | multiple doses: up to Day 1
  The trough concentration observed during the drug administration interval in a steady state (Cmin,ss) after multiple doses
PK parameter AUC0-t | single dose：up to Day 6 ; multiple doses: up to Day 8
  Area under the concentration-time curve (AUC0-t) from time zero to time "t" after single dose and in a steady state after multiple doses
PK parameter AUC0-∞ | single dose：up to Day 6 ; multiple doses: up to Day 8
  AUC from time zero to infinity (AUC0-∞) after single dose and in a steady state after multiple doses
PK parameter AUCtau,ss | multiple doses: up to Day 1
  AUC for the drug administration interval in a steady state (AUCtau,ss) after multiple doses
PK parameter t1/2 | single dose：up to Day 6 ; multiple doses: up to Day 8
  Terminal-phase elimination half-life (t1/2) after single dose and in a steady state after multiple doses

CONTACTS AND LOCATIONS:
Locations (1):
- The Third Xiangya Hospital of Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No